CLINICAL TRIAL: NCT06145568
Title: Maternal & Infant Morbidity and Mortality
Status: Not yet recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Ebony Hilton, Dr. Ebony Hilton, University of Virginia
Other Study IDs: HSR230385
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Preg Complications: Hemorrhagic; Infant, Premature, Diseases; Preg Complications: Hemorrhagic Intervillous of Placenta; Preg Complications: Bleeding From Female Genital Tract; Preg Complic - Malig Hypertension and / or Reason for Care During Childbirth
Keywords: pregnancy complications; hemorrhagic; hypertension; premature infants; bleeding
MeSH Terms: conditions — Infant, Premature, Diseases; Pregnancy Complications; Hypertension; Premature Birth; Hemorrhage

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women: Pregnant Women
  Interventions: Other: Pregnant Women

INTERVENTIONS:
Other: Pregnant Women — We want to quantify Minority Americans at risk of pregnancy complications

SUMMARY:
The purpose of this project is to evaluate maternal and infant outcomes based on race at UVA hospital. Health inequities are influenced by a combination of Social, Political, and Clinical determinants of health. Our hypothesis is that patients with minority status, particularly Black and Hispanic Americans, are more likely to have poor outcomes (based on various health metrics) compared to Non-Black, Non-Hispanic patients. We hypothesize further that it is likely not far off from national trends, which indicate that Black parturients are x4 more likely to die during childbirth, and Black children are 2.4x more likely to die before their first birthday than Non-Hispanic White children.

The EPIC database will be used on an institutional basis to obtain information and accessed by UVA statistician to perform the research described in this submission. The dataset does contain a few direct identifiers of medical record numbers, dates, and postal number. We anticipate that all statistical analysis will be performed at UVA by participating faculty/staff.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate maternal and infant outcomes based on race at UVA hospital. Health inequities are influenced by a combination of Social, Political, and Clinical determinants of health. Our hypothesis is that patients with minority status, particularly Black and Hispanic Americans, are more likely to have poor outcomes (based on various health metrics) compared to Non-Black, Non-Hispanic patients. We hypothesize further that it is likely not far off from national trends, which indicate that Black parturients are x4 more likely to die during childbirth, and Black children are 2.4x more likely to die before their first birthday than Non-Hispanic White children.

The EPIC database will be used on an institutional basis to obtain information and accessed by UVA statistician to perform the research described in this submission. The dataset does contain a few direct identifiers of medical record numbers, dates, and postal number. We anticipate that all statistical analysis will be performed at UVA by participating faculty/staff.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

* N/A

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy complications as a function of minority status | 10 years
  Pregnancy complications as a function of minority status

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris E. US Maternal Mortality Continues to Worsen. JAMA. 2023 Apr 18;329(15):1248. doi: 10.1001/jama.2023.5254. No abstract available. PMID 36988993
- [Background] Himmelstein G, Desmond M. Association of Eviction With Adverse Birth Outcomes Among Women in Georgia, 2000 to 2016. JAMA Pediatr. 2021 May 1;175(5):494-500. doi: 10.1001/jamapediatrics.2020.6550. PMID 33646291
- [Background] Johnson-Agbakwu CE, Ali NS, Oxford CM, Wingo S, Manin E, Coonrod DV. Racism, COVID-19, and Health Inequity in the USA: a Call to Action. J Racial Ethn Health Disparities. 2022 Feb;9(1):52-58. doi: 10.1007/s40615-020-00928-y. Epub 2020 Nov 16. PMID 33197038
- [Background] Boyer BT, Lowell GS, Roehler DR, Quinlan KP. Racial and ethnic disparities of sudden unexpected infant death in large US cities: a descriptive epidemiological study. Inj Epidemiol. 2022 Mar 25;9(1):12. doi: 10.1186/s40621-022-00377-7. PMID 35337375
- See also: Maternal Mortality Rates in the United States, 2021 (cdc.gov) — https://www.cdc.gov/nchs/data/hestat/maternal-mortality/2021/maternal-mortality-rates-2021.htm#fig1